CLINICAL TRIAL: NCT02668029
Title: Effect of Ambulatory Oxygen on the Walking Test in Patients With Pulmonary Fibrosis Normoxemic at Rest Who Desaturate on Exercise
Brief Title: Effect of Ambulatory Oxygen on the Walking Test in Patients With Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Piersante Sestini, associate professor, University of Siena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: WalkO2
Record Dates: First submitted 2016-01-22; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Pulmonary Fibrosis
Keywords: Oxygen therapy
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — Oxygen; Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxygen (Experimental): oxygen administered through a nasal cannula at a personalized, fixed flow
  Interventions: Drug: oxygen
- medical air (Placebo Comparator): Medical air administered through a nasal cannula at the same flow
  Interventions: Drug: medical air

INTERVENTIONS:
Drug: oxygen — information already included in arm/group descriptions.
  Other Names: ambulatory oxygen
  Arms: oxygen
Drug: medical air — Placebo
  Other Names: Placebo
  Arms: medical air

SUMMARY:
Patients with pulmonary fibrosis often desaturate on exercise. There are no data showing whether ambulatory oxygen can be useful to improve exercise capacity in this condition. Ambulatory ambulatory oxygen is often denied to these patients based on studies conducted on patients with chronic obstructive pulmonary disease, a completely different condition for physiopathology, prognosis, and response to therapy. We therefore planned a controlled study to verify the usefulness of ambulatory oxygen in patients with pulmonary fibrosis

DETAILED DESCRIPTION:
Criteria for inclusion: Patients with a diagnosis of pulmonary fibrosis of any kind, with oxygen saturation >90% in ambient air at rest, showing a desaturation <88% during a preliminary 6 minutes walking test Criteria for exclusion: Inability to give consent, age <18 or >85 years, walking problems from causes different from pulmonary disease

Procedure:

In a preliminary session, the flow of oxygen needed to prevent desaturation during walking is established according to a validated protocol Guyatt et al, Am J Respir Crit Care Med 2001,163:,942-946.) Two 6 minutes walking tests are then performed in a corridor, at least 30' apart, during administration of oxygen or medical air, in random order and double blind, at the same pre-determined flow, administered through a nasal cannula connected to a wall outlet (concealed from sight, being in a side rum at about mid distance in the corridor) through a 10 mt plastic tubing. Oxygen saturation and pulse rate are monitored through a dedicated recording oximeter (Minoxy, Cosmed) , whose display is concealed to both the patient and the operator, with an alarm set for oxygen saturation <70%, to stop the test in case severe desaturation would occur Data are then transferred to computer for analysis only after both test are performed. Walked distance is recorded by the operator unaware of treatment.

At the end of each test, a short questionnaire is administered with 10 cm Visual Analogue Scales (VAS) for dyspnoea, fatigue, and preference compared to performing the test without any treatment. At the end of the second test a further scale is submitted, asking about the preference between the two treatments.

Primary outcomes are the distance walked and the difference in preference of the two treatments compared o no treatment. Secondary outcomes are differences in minimal saturation level and maximal pulse rate during the test and in the report of dyspnea and fatigue at the end of the test, and the reported preference between the two treatments.

Statistical analysis to evaluate the effect of the treatment on walking distance, heart frequency and oxygen saturation is performed using generalized linear model with a gaussian family and identity link and including order of treatment as a fixed effect. Parameters evaluated using VAS are analyzed using Koch adaptation of Wilkoxon rank test (Senn SS. Cross-over Trials in Clinical Research, 2nd Edition. Wiley 2002)

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary fibrosis of any cause
* Oxygen saturation => 90% at rest in ambient air, and <88% during walking test

Exclusion Criteria:

* Inability to give consent
* Walking impaired by any condition except pulmonary disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
distance walked | end of test (6 minutes)
  recorded by operator
Difference in preference of the two treatments compared to no treatment. | end of test (6 minutes)
  VAS scale

SECONDARY OUTCOMES:
Difference in oxygen saturation level | Walking test (6 min)
  Digitally recorded
Difference in heart rate | Walking test (6 min)
  Digitally recorded
Difference in dyspnea at the end of test | End of test (6 min)
  VAS
Difference in fatigue at the end of test | End of test (6 min)
  VAS
Preference between the two treatments | End of both tests (45 min)
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: Piersante Sestini, MD, Principal Investigator — University of Siena

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guyatt GH, Nonoyama M, Lacchetti C, Goeree R, McKim D, Heels-Ansdell D, Goldstein R. A randomized trial of strategies for assessing eligibility for long-term domiciliary oxygen therapy. Am J Respir Crit Care Med. 2005 Sep 1;172(5):573-80. doi: 10.1164/rccm.200412-1692OC. Epub 2005 May 18. PMID 15901604
- [Derived] Ciarleglio G, Cameli P, Bennett D, Cekorja B, Rottoli P, Renzoni EA, Sestini P, Bargagli E. Objective Effects and Patient Preferences for Ambulatory Oxygen in Fibrotic Interstitial Lung Disease With Isolated Exertional Hypoxaemia: A Placebo-Controlled 6-Minute Walk Test Study. Respirology. 2025 Jul;30(7):644-651. doi: 10.1111/resp.70020. Epub 2025 Mar 11. PMID 40069946